CLINICAL TRIAL: NCT05404906
Title: Randomized, Multicenter, Phase 3 Study of Azacytidine (AZA) + Venetoclax as Maintenance Therapy in Patients With AML in Remissionin Younger Adults With Favorable-risk AML in First Remission After Conventional Chemotherapy
Brief Title: AZA + Venetoclax as Maintenance Therapy in Younger Adults With AML in First Remission
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ-AML124
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia (AML) in Remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (azacytidine+venetoclax) (Experimental): Participants will receive azacytidine QD, on Days 1-5 and venetoclax QD, on Days 1-14 of each 28-day cycle for 8 cycles.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Other: Supportive care
- Comparator ( best supportive care) (Experimental): Participants will receive observation and supportive care during remission.
  Interventions: Other: Supportive care

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5-Azacytidine
  Arms: Treatment (azacytidine+venetoclax)
Drug: Venetoclax — Given PO
  Other Names: ABT-199; GDC-0199; Venclexta
  Arms: Treatment (azacytidine+venetoclax)
Other: Supportive care — Patients will receive disease monitoring and supportive care for any complication.

SUMMARY:
This phase III trial is conducted to evaluate if azacitidine in combination with venetoclax as maintenance therapy improves relapse-free survival (RFS) for younger adults with favorable-risk acute myeloid leukemia (AML) who remained in first complete remission (CR1) following intensive consolidation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of favorable-risk acute myeloid leukemia (AML) according to revised 2017 European LeukemiaNet genetic risk stratiﬁcation and are not immediate candidates for allogeneic stem cell transplant.
2. Aged 18-64 years.
3. Patients who have received remission induction therapy and 3-4 HiDAC or medium-dose cytarabine-based consolidation and are in their first remission.
4. ECOG performance status of < or = 3.
5. Adequate organ function as follows:

   1. Serum total bilirubin < or = to 3 X the Upper Limit of Normal (ULN)
   2. Aspartate Transaminase and alanine transaminase < or = to 3 x ULN
   3. Ccr（Creatinine Clearance Rate) > or ＝60 ml/min
   4. Left ventricular ejection fraction > or ＝50% determined by ultrasound.
6. For females of childbearing age, they should have a negative serum or urine pregnancy test within 10 to 14 days of enrolling.
7. For males of childbearing age, they should take effective contraceptive methods throughout the treatment period and up to 30 days after discontinuing treatment.
8. Ability to understand and sign informed consent.

Exclusion Criteria:

1. Acute promyeloid leukemia.
2. Patients with active central nervous system (CNS) leukemia.
3. Previously diagnosed with myelodysplastic syndrome (MDS) or myeloproliferative neoplasm(MPN) and progressed to AML.
4. Patients with other progressive malignancies.
5. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to uncontrolled and/or active systemic infection (viral, bacterial or fungal).
6. Patients who have participated in other trials within 30 days before signing the informed consent.
7. Females who are pregnant or lactating or intending to become pregnant during the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | From date of complete remission (CR) or complete remission with incomplete count recovery (CRi), to relapse or death from any cause, up to approximately 3 years
  RFS is defined as the number of days from CR/CRi to the date of relapse or the date of death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve Minimal Minimal Residual Disease (MRD) Negative Conversion | Measured From Baseline to approximately 3 years
  The MRD conversion rate is defined as the percentage of participants deemed MRD positive (≥ 10^-3) at study initiation who converted to MRD of < 10^-3 in the bone marrow after randomization or initiation of treatment.
Complete remission duration (CRd) | From date of CR/CRi to approximately 3 years
  CRd is defined as time from CR/CRi until date of confirmed relapse
Overall Survival (OS) | Time from treatment to death from any cause, up to approximately 3 years
  OS is defined as the number of days from the date of study treatment to the date of death.
Event free survival (EFS) | Time from treatment to relapse，withdrawal from study due to adverse event and death from any cause, up to approximately 3 years
  EFS is defined as time from the start of study treatment until date of first confirmed relapse, withdrawal from study due to adverse event, or death due to any cause,
Incidence of adverse events | Time from treatment to approximately 3 years
  The NCI Common Toxicity Criteria (CTCAE 5.0) is used to grade adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, Principal Investigator — First Affiliated Hospital of Soochow University
Locations (2):
- China (2):
  - First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No